CLINICAL TRIAL: NCT05563740
Title: Assisted vs Unassisted Domiciliary Alcohol Detoxification: A Randomised Control Trial
Brief Title: Psychosocial Intervention For Domiciliary Alcohol Detoxification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Sneha B Suresh (Other)
Responsible Party: Sponsor-Investigator, Dr Sneha B Suresh, Principle Investigator, Goa Medical College
Organization: Goa Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GMC121019
Record Dates: First submitted 2022-09-23; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol withdrawal; Home detoxification; Domiciliary Detoxification
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): All received care for alcohol withdrawal state as is routinely provided at the centre by their respective treating doctors and followed up as directed. All treatment and follow up decisions were made by the respective treating doctors. Study team did not have any role in it.
  In addition all received a session of Brief Intervention (BI) for alcohol, at the time of recruitment and again after completing detoxification. Further, patient or designated caregiver received daily phone calls and Information was provided regarding any queries related to their withdrawal or detoxification process. Adverse outcomes such as sedation, seizure, confusion were enquired for and records were kept. Patient was encouraged to continue the treatment and report back for scheduled follow ups and in case of any adverse outcomes patient was asked to report back to the treating doctor and an appointment was facilitated. Phone calls were discontinued once detoxification (CIWA < 8) was complete.
  Interventions: Other: Psychosocial
- Control Group (No Intervention): All participants received care for alcohol withdrawal state as is routinely provided at the centre by their respective treating doctors and followed up as directed. All treatment and follow up decisions were made by the respective treating doctors. Study team did not have any role in it.

INTERVENTIONS:
Other: Psychosocial — Daily telephone calls with two sessions of Brief Interventions for alcohol
  Arms: Intervention Group

SUMMARY:
Alcohol Use Disorders (AUD) form a major public health issue in India. In a densely populated country with limited mental health resources, it is challenging to treat those with AUD appropriately. Detoxification is the first step in dealing with clinically significant AUD. Institution based detoxification is not universally available and home based detoxification is mired with poor outcomes with people resuming drinking behaviour. This trail therefore aimed to study the effect of a psychosocial intervention to improve the outcome of domiciliary alcohol detoxification. The intervention involved Brief Interventions for alcohol and daily telephone monitoring and psychosocial support of patients undergoing home detoxification.

DETAILED DESCRIPTION:
Background: Alcohol use is a major contributor to the worldwide disease burden. Alcohol consumption has dropped in high-income nations over the last decade, whereas it has increased in some low- and middle-income countries in Southeast Asia, including India, where alcohol use resulted in 3.4 million deaths and 14.7 million disability-adjusted life years for the year 2019.

According to World Health Organization (WHO) estimates, total adult alcohol per capita consumption (APC, in liters of pure alcohol) in India has rapidly increased from 2.3 liters (2000) to 5.5 liters (2018), with further rises anticipated until 2025, thus making alcohol use disorders an important public health issue which needs urgent attention from all stakeholders.

A considerable proportion of persons in India with Alcohol Use Disorder (AUD) do not have access to treatment for their alcohol-related disorders, resulting in an 86 percent treatment gap. Community based care options being limited; treatment for AUD is largely dependent upon institutional care, which is both limited and strained. AUD encompasses a broad range of drinking behaviors, however for the purpose of this study the term AUD will refer to drinking behavior needing clinical attention.

Detoxification is the initial stage in therapy for AUD. It can take place in the community or in an inpatient facility; the option is based on the degree of the alcohol use. Evidence suggests that community detoxification is preferable to inpatient detoxification in terms of overall success, cost-effectiveness, feasibility, treatment gap reduction, and client acceptability.

Domiciliary alcohol detoxification is a process where the management of detoxification is advised at the level of patient's home, where an alcohol dependent patient is safely detoxified without admission to an inpatient unit. Whereas in assisted domiciliary alcohol detoxification additional monitoring is provided while the patient undergoes detoxification in the community. The implementation of Mental Health Care Act 2017 recommends treatment of the patient in the community, thus domiciliary detoxification is a step in that direction.

The aim of this study was to trail an intervention that assisted a randomly assigned group of patients undergoing domiciliary detoxification. The assistance was through daily phone call monitoring until successful detoxification with brief intervention sessions on two occasions; with the outcome measured as successful detoxification and abstinence at the end of one month.

Methodology:

Study setting: This study was based at the out-patient department of a tertiary care psychiatry hospital in Goa, India.

Study Design: Randomised Control Trial Sample and sample size: 100 consenting male patients aged between 18-65 years who presented in alcohol withdrawal state and were advised Domiciliary Detoxification by treating doctor were included in the study. The sample size was a pragmatic estimate based on feasibility.

Procedure: Eligible patients were approached and written consent was obtained after detailed explanation of the study. Baseline assessment of all participants was done using a) Severity of Alcohol Dependence Questionnaire (SAD-Q) for severity of alcohol dependence. The SAD-Q has been extensively used in a number of studies in India b) Readiness to Change Questionnaire, treatment version (RCQ-TV) for motivation to quit alcohol. This scale is based on Prochaska and DiClemente's stages of change model, for assignment of excessive drinkers to Precontemplation, Contemplation, and Action stages. Researchers throughout the world have used this questionnaire as a simple mean to assess the stage of motivation of an individual and c) Clinical Institute Withdrawal Assessment of Alcohol scale, Revised (CIWA-Ar) for severity of withdrawal. A cut-off of 8 was considered for intake as scores below 8 usually do not need medical management. A vernacular version of the scales was generated using the translation-back translation method. Predesigned semi-structured questionnaire was used to assess the socio-demographic variables and drinking related variables.

Randomisation: Following baseline assessment, randomisation was carried out using pre-randomised and sealed envelopes to assign the subject either into intervention or control group. Randomisation was done by third party not involved in any way with the study. No blinding could be carried out as it was a single investigator study however steps to avoid bias were taken by doing the baseline assessment prior to randomisation.

Both groups (Intervention and Control) received care for alcohol withdrawal state as is routinely provided at the centre by their respective treating doctors and followed up as directed. All treatment and follow up decisions were made by the respective treating doctors. Study team did not have any role in it.

Intervention: The intervention group in addition received a session (approx. 15 min) of Brief Intervention (BI) for alcohol, at the time of recruitment and again after completing detoxification. The BI session was delivered on structured lines based on psychoeducation and personalised feedback. It focussed on making patient aware of the potential harm if alcohol was continued, mainly in terms of medical, social, financial aspects and encouraged abstinence. BI model was selected to keep the intervention simple and feasible. Further, patient or designated caregiver received daily phone calls and Information was provided regarding any queries related to their withdrawal or detoxification process. Adverse outcomes such as sedation, seizure, confusion were enquired for and records were kept. Patient was encouraged to continue the treatment and report back for scheduled follow ups and in case of any adverse outcomes patient was asked to report back to the treating doctor and an appointment was facilitated. Phone calls were discontinued once detoxification (CIWA < 8) was complete.

Outcome assessment: Outcome measurement for successful detoxification was done at every follow up for both groups. A CIWA score of less than 8 was considered as successful completion of detoxification. Similarly, outcome assessment for abstinence at one month was done using the Time Line Follow Back Method after one month of detoxification either in person or by phone call. The Alcohol TLFB is a drinking assessment method that obtains estimates of daily drinking. People give retrospective estimates of their daily drinking over a specified time period that can vary up to 12 months from the interview date using a calendar. This method has been used across wide settings.

Data analysis and interpretation: Data was analysed using the Statistical Package for Social Sciences (SPSS) for Windows software (version 22.0; SPSS Inc., Chicago). Descriptive statistics such as mean and standard deviation (SD) for continuous variables and frequencies and percentages for categorical Variables were calculated. Association between study group and other categorical variables were analysed using chi-square test of independence and unpaired t-test for continuous variables. Level of significance was set at p<0.05.

Ethical considerations: The study received ethical clearance from the Institutional Ethics Committee at The Goa Medical College, Goa. Written Informed consent was obtained after thorough description of the study to the participants in their own vernacular. All data was kept confidential and privacy was ensured. All relevant information was shared with the treating doctor with consent of the patient. Patients in the control group received the same care as is routinely provided at the hospital. Those patients who had resumed drinking at the end of the trial period received brief counselling regarding drinking and were directed to visit for further assistance.

ELIGIBILITY:
Inclusion Criteria: Consenting male patients aged between 18-65 years who presented in alcohol withdrawal state and were advised Domiciliary Detoxification by treating doctor.

-

Exclusion Criteria:

* Nil

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Succesful Detoxification | Up to four weeks
  Proportion of participants successfully completing detoxification as indicated by CIWA score of less than 8

SECONDARY OUTCOMES:
Abstinence at one month | One month
  Total duration in days abstinent from alcohol at one month from detoxification measured on Time Line Follow Back method.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Rane, Principal Investigator — IPHB
Locations (1):
- Institue of Psychiatry & Human Behaviour, Bambolim, Goa, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manthey J, Shield KD, Rylett M, Hasan OSM, Probst C, Rehm J. Global alcohol exposure between 1990 and 2017 and forecasts until 2030: a modelling study. Lancet. 2019 Jun 22;393(10190):2493-2502. doi: 10.1016/S0140-6736(18)32744-2. Epub 2019 May 7. PMID 31076174
- [Background] National Collaborating Centre for Mental Health (UK). Alcohol-Use Disorders: Diagnosis, Assessment and Management of Harmful Drinking and Alcohol Dependence. Leicester (UK): British Psychological Society (UK); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK65487/ PMID 22624177
- [Background] GBD 2016 Risk Factors Collaborators. Global, regional, and national comparative risk assessment of 84 behavioural, environmental and occupational, and metabolic risks or clusters of risks, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1345-1422. doi: 10.1016/S0140-6736(17)32366-8. PMID 28919119
- [Background] 4. Hammer JH, Parent MC, Spiker DA, World Health Organization. Global status report on alcohol and health 2018 [Internet]. Vol. 65, Global status report on alcohol. 2018. 74-85 p. Available from: http://www.who.int/substance_abuse/publications/global_alcohol_report/msbgsruprofiles.pdf%0Ahttp://www.ncbi.nlm.nih.gov/pubmed/29355346
- [Background] Rastogi A, Manthey J, Wiemker V, Probst C. Alcohol consumption in India: a systematic review and modelling study for sub-national estimates of drinking patterns. Addiction. 2022 Jul;117(7):1871-1886. doi: 10.1111/add.15777. Epub 2022 Jan 10. PMID 34873774
- [Background] Nadkarni A, Velleman R, Bhatia U, Fernandes G, D'souza E, Murthy P. Home-detoxification and relapse prevention for alcohol dependence in low resource settings: An exploratory study from Goa, India. Alcohol. 2020 Feb;82:103-112. doi: 10.1016/j.alcohol.2019.08.006. Epub 2019 Aug 29. PMID 31473304
- [Background] Nemlekar S, Gaonkar P, Rane A. Domiciliary alcohol detoxification outcomes: a study from Goa, India. J Addict Dis. 2021 Jan-Mar;39(1):105-108. doi: 10.1080/10550887.2020.1826103. Epub 2020 Oct 20. PMID 33079007
- [Background] 8. The Mental Health Care Act 2017. Available from: http://www.prsindia.org/uploads/media/Mental%20Health/Mental%20Healthcare%20Act,%202017.pdf
- [Background] D'Souza PC, Mathai PJ. Motivation to change and factors influencing motivation in alcohol dependence syndrome in a tertiary care hospital. Indian J Psychiatry. 2017 Apr-Jun;59(2):183-188. doi: 10.4103/psychiatry.IndianJPsychiatry_262_15. PMID 28827865
- [Background] Johnson PR, Britto C, Sudevan KJ, Bosco A, Sreedaran P, Ashok MV. Resilience in Wives of persons with Alcoholism: An Indian exploration. Indian J Psychiatry. 2018 Jan-Mar;60(1):84-89. doi: 10.4103/psychiatry.IndianJPsychiatry_271_14. PMID 29736068
- [Background] Baby S, Murthy P, Thennarasu K, Chand PK, Viswanath B. Comparative outcome in patients with delirium tremens receiving care in emergency services only versus those receiving comprehensive inpatient care. Indian J Psychiatry. 2017 Jul-Sep;59(3):293-299. doi: 10.4103/psychiatry.IndianJPsychiatry_260_17. PMID 29085087
- [Background] Gupta A, Murthy P, Rao S. Brief screening for cognitive impairment in addictive disorders. Indian J Psychiatry. 2018 Feb;60(Suppl 4):S451-S456. doi: 10.4103/psychiatry.IndianJPsychiatry_41_18. PMID 29540913
- [Background] Gulati P, Chavan BS, Sidana A. Authors' reply to commentary on "Gulati P, Chavan BS, Sidana A. Comparative efficacy of baclofen and lorazepam in the treatment of alcohol withdrawal syndrome". Indian J Psychiatry. 2019 Nov-Dec;61(6):652-653. doi: 10.4103/psychiatry.IndianJPsychiatry_325_19. No abstract available. PMID 31896877
- [Background] Sullivan JT, Sykora K, Schneiderman J, Naranjo CA, Sellers EM. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar). Br J Addict. 1989 Nov;84(11):1353-7. doi: 10.1111/j.1360-0443.1989.tb00737.x. PMID 2597811
- [Background] Prochaska JO, Velicer WF. The transtheoretical model of health behavior change. Am J Health Promot. 1997 Sep-Oct;12(1):38-48. doi: 10.4278/0890-1171-12.1.38. PMID 10170434
- [Background] 18. Waters AF. Readiness to change and smoking expectancies among adult male substance users currently in substance use treatment by. 2020;(December).
- [Background] Timko C, Below M, Schultz NR, Brief D, Cucciare MA. Patient and program factors that bridge the detoxification-treatment gap: a structured evidence review. J Subst Abuse Treat. 2015 May;52:31-9. doi: 10.1016/j.jsat.2014.11.009. Epub 2014 Dec 3. PMID 25530425
- [Background] Sarkar S, Pakhre A, Murthy P, Bhuyan D. Brief Interventions for Substance Use Disorders. Indian J Psychiatry. 2020 Jan;62(Suppl 2):S290-S298. doi: 10.4103/psychiatry.IndianJPsychiatry_778_19. Epub 2020 Jan 17. No abstract available. PMID 32055071
- [Background] Hjorthoj CR, Hjorthoj AR, Nordentoft M. Validity of Timeline Follow-Back for self-reported use of cannabis and other illicit substances--systematic review and meta-analysis. Addict Behav. 2012 Mar;37(3):225-33. doi: 10.1016/j.addbeh.2011.11.025. Epub 2011 Nov 26. PMID 22143002